CLINICAL TRIAL: NCT02879773
Title: An Observational Study of Non Contrast Computed Tomography in Assessment of Regional Ventilation of the Lung.
Brief Title: Computed Tomography Assessment of Regional Ventilation (CURVE)
Acronym: CURVE
Status: Completed | Type: Observational
Sponsor: Heart of England NHS Trust (Other)
Collaborators: British Lung Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 178070
Record Dates: First submitted 2016-08-05; First posted 2016-08-26 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Lung Neoplasms; Emphysema; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive
Keywords: Respiratory Function Tests; Computed tomography; Thoracic surgical procedures; Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Emphysema; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lung cancer: Patients undergoing thoracic surgery for suspected or confirmed lung cancer; including wedge resection, segmentectomy, lobectomy, bilobectomy or pneumonectomy. CTPVe will be modelled to predict postoperative lung function.
  Interventions: Radiation: CTPVe
- Emphysema: Patients undergoing assessment of emphysema/chronic obstructive pulmonary disease (COPD) for potential surgical intervention; including lung volume reduction surgery, endobronchial valve insertion or endobronchial coil insertion. CTPVe will be modelled to predict postoperative lung function.
  Interventions: Radiation: CTPVe
- Interstitial lung disease: Patients undergoing assessment or treatment of suspected or confirmed interstitial lung disease. CTPVe will be modelled to aid diagnosis of the subtype of interstitial lung disease confirmed by histological diagnosis.
  Interventions: Radiation: CTPVe

INTERVENTIONS:
Radiation: CTPVe — Non contrast computed tomography (CTPVe) scan during end inspiration and end expiration in supine position

SUMMARY:
This study uses CT scans to assess airflow in the lung, the scan is quick, cheap and painless. The information from the scan may help doctors tell which patients are suitable to have surgery to cure early stage lung cancer. It may also help doctors tell which patients would benefit from surgery for emphysema and diagnose types of lung disease. The investigators will follow up patients who go through surgery to test how well the scan predicts the function of the lung after surgery. The investigators will follow patients being investigated for lung disease to test how accurate the scan is at the getting the diagnosis right.

DETAILED DESCRIPTION:
CT scans during breathing in and breathing out (CTPVe) can assess regional airflow within the lung, using newly developed software as described by Aliverti et al. This provides information about the function of each part of the lung. The investigators aim to assess the feasibility of a larger trial using CTPVe to guide treatment of lung diseases and develop the statistical models needed for use in these trials.

Surgery provides the best prospect of a cure in early Non-small cell lung cancer. In the UK only half of people with early lung cancer undergo surgery and poor lung function may be a barrier to removal of part of the lung. Many patients with lung cancer also have emphysema or other lung diseases that reduce lung function. Actual post-operative lung function is often better predicted by current methods. The investigators will assess regional airflow in the lung and compare the airflow to the patients lung function both before and after surgery to assess if CTPVe can predict postoperative lung function, enabling more people to be considered suitable for curative surgery,

Severe emphysema is debilitating, some surgical treatments can improve the symptoms of emphysema; these include lung volume reduction surgery, endobronchial valves and endobronchial coils. Each of these are only suitable for certain patients and it is difficult to predict who will benefit most. The investigators will assess regional airflow in the lung and compare the airflow to the patients lung function before and after these treatments for emphysema to assess if CTPVe can predict who will benefit from surgery.

There are hundreds of subtypes of interstitial lung disease that respond to different types of treatment but diagnosing the subtype can be very difficult. Patients may need to undergo surgery to get the diagnosis of their subtype and this is associated with major risks, including death. The investigators will assess the regional airflow in the lung and compare the pattern to the final subtype of interstitial lung disease to assess if CTPVe could mean future patients do not need surgery for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Undergoing assessment or treatment of parenchymal lung disease which involves CT scanning
* Able to understand the study information and provide written informed consent

Exclusion Criteria:

* Pregnancy
* Inability to follow breath hold instructions for CT scan
* Body size exceeding the capacity of CT scanner
* Previous chest wall resection
* Presence of implantable device that would cause artefacts on CT images including ICD, pacemaker, internal fixation of rib fracture, ventricular assist device, spinal rods/pedicle screws, shoulder replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adults being assessed or treated in a hospital with a patient case mix and size typical of thoracic practice in England. As a tertiary referral centre patients will come from a wide geographical range and from both rural and urban settings.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible patients screened who consent to participate | 2 years

SECONDARY OUTCOMES:
Change in gas transfer | 3-6 months
  Change in gas transfer factor (DLCO) reported as percentage of predicted value.
Change in FEV1 | 3-6 months
  Change in forced expiratory volume in 1 second reported as percentage of predicted value.
Diagnosis | 3-6 months
  The histological or multidisciplinary team consensus diagnosis of subtype of interstitial lung disease (if applicable)
Change in perception of breathlessness | 3-6 months
  Change in the patient perception of breathlessness measured suing Borg scale 0-10
Regional ventilation | 3-6 months
  Regional ventilation of the lung as assessed on CTPVe scanning, reported in millilitres of air per gram of lung tissue
Percentage of patients who gave consent to participate but were later withdrawn | 2 years
Number of patients recruited per month | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Babu Naidu, MBBS, Principal Investigator — Heart of England NHS Foundation Trust
Locations (1):
- Heart of England NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aliverti A, Pennati F, Salito C, Woods JC. Regional lung function and heterogeneity of specific gas volume in healthy and emphysematous subjects. Eur Respir J. 2013 May;41(5):1179-88. doi: 10.1183/09031936.00050112. Epub 2012 Aug 9. PMID 22878884